CLINICAL TRIAL: NCT03502798
Title: Coherence Imaging of the Cervical Epithelium With Scanning a/LCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Jacobi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00070555_1; R01CA167421 (NIH)
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Cervical Dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- scanning a/LCI (Experimental)
  Interventions: Device: scanning a/LCI

INTERVENTIONS:
Device: scanning a/LCI — Imaging of the cervical epithelium using the scanning a/LCI device.

SUMMARY:
The purpose of this study is to develop a low coherence interferometry (LCI) endoscopic probe that can examine the cervix for evidence of cervical dysplasia. The device will make optical measurements of the cervix to determine:

1. the difference between two different types of cervical cells: ectocervical cells and endocervical cells. Cervical dysplasia is most likely to occur at the junction between these two types of cells.
2. features of individual cervical cells that indicate whether the cell is normal or abnormal (cervical dysplasia).

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* willing to abstain from sexual intercourse for at least 24 hours before study visit

Exclusion Criteria:

* pregnant
* have a current gynecological infection or discharge
* have had any cervical surgery
* had medical or cosmetic surgery involving the reproductive organs or genitals within the past 6 months
* currently enrolled in any research studies involving the application of vaginal formulations
* employed or supervised by the study investigators
* have any other condition, that, in the opinion of the study clinician, would contraindicate participation in the study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wax, Ph.D., Principal Investigator — professor
Locations (2):
- United States (2):
  - Jacobi Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Scanning a/LCI (Pilot): Pilot study conducted at Duke University (Durham, NC). Exclusion criteria included: current gynecological infection or discharge, prior cervical surgery, or positive urine pregnancy test. The scanning a/LCI probe was inserted into the vagina and placed against the cervix using direct visualization provided by a white light camera incorporated into the probe. Optical interferometric data were acquired to characterize the instrument's ability to detect cervical dysplasia via depth-resolved nuclear morphology measurements.
- Scanning a/LCI (Jacobi): Primary arm of present study, conducted at New York City Health + Hospitals / Jacobi (Bronx, New York, NY). Exclusion criteria included: current gynecological infection or discharge, prior cervical surgery, or positive urine pregnancy test. In addition, participants abstained from sexual intercourse for at least 24 hours prior to the study visit.
  A speculum was inserted prior to the a/LCI probe for ease of tissue biopsy collection after a/LCI scanning. The scanning a/LCI probe was inserted through speculum and placed against the cervix using white light visual guidance from the probe's integrated camera. The a/LCI imaging sequence was initiated, with 36 scan points spaced across an area of 50 mm2. 80 a/LCI optical biopsy scans were at 4 selected biopsy sites (20 per quadrant). The a/LCI probe was removed and a Wallach colposcope was used to take a digital image of the cervix for co-registration with the a/LCI image. Some women underwent a previously scheduled loop electrosurgical excision procedure (LEEP) immediately following data collection; tissue biopsies were taken either with the assistance of the colposcope or during the LEEP and all specimens were analyzed by pathologists to provide a histological diagnosis for comparison with the a/LCI measurements. Tissue biopsies for each quadrant were assigned a classification (negative, CIN-1, CIN-2, or CIN-3) as well as notes for any additional findings (koilocytic atypia, abnormal acetowhite epithelium, etc.).
Period: Overall Study
Arm/Group | Scanning a/LCI (Pilot) | Scanning a/LCI (Jacobi)
Started | 5 | 40
Completed | 5 | 33
Not Completed | 0 | 7
Not completed — equipment failure | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scanning a/LCI (Pilot) | Scanning a/LCI (Jacobi) | Total
Number analyzed (Participants) | 5 | 40 | 45
Age, Continuous [Mean (Full Range); unit: years] — Population: Age was not recorded for 2 participants in the Jacobi arm.
  years
    number analyzed (Participants) | 5 | 38 | 43
    (all) | 26 [21 to 34] | 35 [23 to 49] | 34 [21 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 40 | 45
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 23 | 23
  Not Hispanic or Latino | 5 | 14 | 19
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 11 | 13
  White | 2 | 17 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 11 | 11

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Scanning a/LCI Probe to Detect Cervical Dysplasia as Measured by Percentage of Correctly Identified Positive Biopsies
Description: Sensitivity of the scanning a/LCI probe's ability to detect cervical dysplasia determined by calculating the percentage of correctly identified positive optical biopsies measured by the scanning a/LCI probe when compared to the gold standard, histopathology.
  There are two dichotomies of classification used in this study: one that focuses on the morphological differences between cells (histology-based classification), and one that focuses on the urgency of corresponding treatment (response-based classification). In the histology-based classification, a result of benign alone is a negative result and a result of LSIL (low-grade squamous intraepithelial lesion) or HSIL (high-grade squamous epithelial lesion) is a positive result. In the response-based classification, both benign and LSIL are treated as negative results and HSIL is treated as a positive result.
Time Frame: baseline
Population: 40 women enrolled at the Jacobi site, but successful a/LCI scans were only acquired from 20 participants due to equipment failures (mechanical breaks in probe, electrical component failures, software errors). For each participant analyzed, optical biopsies (a/LCI scans) and corresponding physical tissue biopsies were collected at four sites (12, 3, 6, and 9 o'clock). No pilot study participants were analyzed as no physical tissue biopsies were done in the pilot phase.
Measure: Number (95% Confidence Interval); unit: percentage of correct identifications
Units Other Than Participants: biopsies
Arm/Group | Scanning a/LCI (Pilot) | Scanning a/LCI (Jacobi)
Number analyzed (Participants) | 0 | 20
Number analyzed (biopsies) | 0 | 80
percentage of correct identifications
  histology-based classification |  | 90.3 [74.2 to 98.0]
  response-based classification |  | 100.0 [73.5 to 100.0]

2. Primary Outcome: Specificity of Scanning a/LCI Probe to Detect Cervical Dysplasia as Measured by Percentage of Correctly Identified Negative Optical Biopsies
Description: Specificity of the scanning a/LCI probe's ability to detect cervical dysplasia determined by calculating the percentage of correctly identified negative optical biopsies measured by the scanning a/LCI probe when compared to the gold standard, histopathology.
  There are two dichotomies of classification used in this study: one that focuses on the morphological differences between cells (histology-based classification), and one that focuses on the urgency of corresponding treatment (response-based classification). In the histology-based classification, a result of benign alone is a negative result and a result of LSIL (low-grade squamous intraepithelial lesion) or HSIL (high-grade squamous intraepithelial lesion) is a positive result. In the response-based classification, both benign and LSIL are treated as negative results and HSIL is treated as a positive result.
Time Frame: baseline
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of correct identifications
Units Other Than Participants: biopsies
Arm/Group | Scanning a/LCI (Pilot) | Scanning a/LCI (Jacobi)
Number analyzed (Participants) | 0 | 20
Number analyzed (biopsies) | 0 | 80
percentage of correct identifications
  histology-based classification |  | 81.6 [68.0 to 91.2]
  response-based classification |  | 70.6 [58.3 to 81.0]

3. Secondary Outcome: Identification of T-zone by Scanning a/LCI Probe
Description: Ability of scanning a/LCI probe to correctly identify transformation zone (T-zone) compared to colpophotography
Time Frame: baseline
Population: Data not collected due to frequent instrument repairs.
Arm/Group | Scanning a/LCI (Pilot) | Scanning a/LCI (Jacobi)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day of study only
Arm/Group | Scanning a/LCI (Pilot) | Scanning a/LCI (Jacobi)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/40
Other Adverse Events (participants affected / at risk) | 0/5 | 0/40

LIMITATIONS AND CAVEATS:
The fragility of the instrument resulted in repeated breakage. Traveling from Durham to NYC to retrieve the broken instrument, repair it, and send it back several times set the timeline back substantially, resulting in insufficient time to perform the secondary outcome measure.

Instrument fragility, complexity of instrument set up and initiation, and poor signal quality are responsible for the low yield of evaluable a/LCI scans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT03502798/Prot_SAP_000.pdf